CLINICAL TRIAL: NCT02755909
Title: The Effect of Pre-anesthetic Education on Patients' Anxiety Level Undergoing Cardiac Surgery
Brief Title: The Effect of Pre-anesthetic Education on Cardiac Surgery Patients' Anxiety Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Arif H. M. Marsaban, Consultant, Anesthesiologist, Indonesia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes002
Record Dates: First submitted 2016-04-28; First posted 2016-04-29 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Cardiac Surgery Patients
Keywords: Cardiac surgery, anxiety, education
MeSH Terms: conditions — Anxiety Disorders

ARMS (1):
- Subjects (Other): Pra-anesthetic education given to the subjects includes the anatomy of a normal heart, normal blood circulation, anatomy and pathophysiology of the disease in the respected subject, surgery procedures needed, anesthetic procedures needed for the surgery, and cardiopulmonary bypass procedures. Education and discussion were given repeatedly until subjects could repeat the materials given correctly.
  Interventions: Behavioral: Pre-anesthetic Education

INTERVENTIONS:
Behavioral: Pre-anesthetic Education — Education was done before the anesthetic procedure, using a flip chart made by the researchers.

SUMMARY:
The study aims to investigate the effect of pre-anesthetic education on patients undergoing cardiac surgery

DETAILED DESCRIPTION:
Approval from Ethical Committee of Faculty of Medicine University of Indonesia was acquired prior conducting the study. Subjects were given informed consent before enrolling the study. Subjects identification was done using identification form, medical record, Mini Mental State Evaluation (MMSE) and Internal Classification of Diseases (ICD) 10. Subjects' anxiety level were measured using Amsterdam Preoperative Anxiety and Information Scale (APAIS) with the help of the researcher to explain the questions. Then, education were given to the subjects, guided by a flow chart made by the researcher, using verbal and emphatic non-verbal language. If during education subjects got anxious with or without cardiovascular emergencies, education would be stopped, subjects would be eased down. Subject's family would be called in. If the subjects agreed to continue, the study would be carried on, otherwise subjects were dropped out. Benzodiazepin and midazolam 0.5 mg/kgBW would be considered and consulted to a psychiatrist. On the day after the education and discussion, subjects filled in APAIS again before entering the operation room. APAIS score recorded before and after anesthesia would be presented in the means, and analyzed by SPSS using paired T-test (or Wilcoxon test as the alternative test).

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18-65 years old
* Subjects able to read and write properly
* Subjects have adequate communication ability
* Subjects were able to speak Indonesian language properly
* Subjects were planned to undergo cardiac surgery
* Subjects have given informed consent for the anesthetical and surgical procedures.

Exclusion Criteria:

* Subjects who did not give informed consent
* Subjects who had done a cardiac surgery before this study commenced,
* Subjects who had a cognitive/psychiatric problem that decreased communication ability
* Subjects in antianxiety and/or antidepressant treatment.

Drop out criteria:

* Subjects who had anxiety sign and symptoms with/without cardiovascular alarming signs and could not be eased down during education
* Subjects decided to drop out the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Subjects' Anxiety Level before Education | 2 months
  Subjects' anxiety level before education was measure using APAIS instrument.
Subjects' Anxiety Level after Education | 2 months
  Subjects' anxiety level after education was measure using APAIS instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Arif HM Marsaban, Consultant, Principal Investigator — Indonesia University

REFERENCES:
- [Background] Domar AD, Everett LL, Keller MG. Preoperative anxiety: is it a predictable entity? Anesth Analg. 1989 Dec;69(6):763-7. PMID 2589657
- [Background] Maranets I, Kain ZN. Preoperative anxiety and intraoperative anesthetic requirements. Anesth Analg. 1999 Dec;89(6):1346-51. doi: 10.1097/00000539-199912000-00003. PMID 10589606
- [Background] Kiyohara LY, Kayano LK, Oliveira LM, Yamamoto MU, Inagaki MM, Ogawa NY, Gonzales PE, Mandelbaum R, Okubo ST, Watanuki T, Vieira JE. Surgery information reduces anxiety in the pre-operative period. Rev Hosp Clin Fac Med Sao Paulo. 2004 Apr;59(2):51-6. doi: 10.1590/s0041-87812004000200001. Epub 2004 Apr 26. PMID 15122417
- [Background] Valenzuela Millan J, Barrera Serrano JR, Ornelas Aguirre JM. Anxiety in preoperative anesthetic procedures. Cir Cir. 2010 Mar-Apr;78(2):147-51. English, Spanish. PMID 20478116
- [Background] Moerman N, van Dam FS, Muller MJ, Oosting H. The Amsterdam Preoperative Anxiety and Information Scale (APAIS). Anesth Analg. 1996 Mar;82(3):445-51. doi: 10.1097/00000539-199603000-00002. PMID 8623940
- [Background] Wetsch WA, Pircher I, Lederer W, Kinzl JF, Traweger C, Heinz-Erian P, Benzer A. Preoperative stress and anxiety in day-care patients and inpatients undergoing fast-track surgery. Br J Anaesth. 2009 Aug;103(2):199-205. doi: 10.1093/bja/aep136. Epub 2009 May 30. PMID 19483203
- [Background] Laufenberg-Feldmann R, Kappis B. Assessing preoperative anxiety using a questionnaire and clinical rating: a prospective observational study. Eur J Anaesthesiol. 2013 Dec;30(12):758-63. doi: 10.1097/EJA.0b013e3283631751. PMID 23787971
- [Background] Kindler CH, Harms C, Amsler F, Ihde-Scholl T, Scheidegger D. The visual analog scale allows effective measurement of preoperative anxiety and detection of patients' anesthetic concerns. Anesth Analg. 2000 Mar;90(3):706-12. doi: 10.1097/00000539-200003000-00036. PMID 10702461
- [Background] Millar K, Jelicic M, Bonke B, Asbury AJ. Assessment of preoperative anxiety: comparison of measures in patients awaiting surgery for breast cancer. Br J Anaesth. 1995 Feb;74(2):180-3. doi: 10.1093/bja/74.2.180. PMID 7696068
- [Background] Julian LJ. Measures of anxiety: State-Trait Anxiety Inventory (STAI), Beck Anxiety Inventory (BAI), and Hospital Anxiety and Depression Scale-Anxiety (HADS-A). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S467-72. doi: 10.1002/acr.20561. No abstract available. PMID 22588767
- [Background] Bonnet C, Greffier A. Paediatric cardiac catheterization: an information sheet. Arch Cardiovasc Dis. 2013 Apr;106(4):228-37. doi: 10.1016/j.acvd.2013.01.007. Epub 2013 Apr 23. PMID 23706369
- [Background] Bensing J. Doctor-patient communication and the quality of care. Soc Sci Med. 1991;32(11):1301-10. doi: 10.1016/0277-9536(91)90047-g. PMID 2068614